CLINICAL TRIAL: NCT02834741
Title: A Randomized, Double-Blind, Sponsor-Open, Placebo-Controlled, Single and Multiple Ascending Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of Daily Oral NYX2925 in Healthy Volunteers
Brief Title: Safety, Tolerability, PK of Oral NYX-2925 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aptinyx (Industry)
Collaborators: Spaulding Clinical Research LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NYX-2925-1001
Record Dates: First submitted 2016-07-13; First posted 2016-07-15 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — NYX-2925

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SAD Phase (Placebo Comparator): Up to 36 subjects: 50 - 1200 mg NYX-2925, Up to 12 subjects: placebo
  6 additional subjects will receive a fed dose of NYX-2925, 2 additional subjects will receive a fed dose of placebo (Food Effect Cohort)
  6 additional subjects will receive 1 dose of 50 mg NYX-2925 followed by a lumbar puncture at 1 and 4 (3 subjects) or 2 and 8 (3 subjects) hours post dose
  Interventions: Drug: NYX-2925
- MAD Phase (Placebo Comparator): Up to 24 subjects : 150 - 600 mg NYX-2925 daily for 7 days, up to 6 subjects : placebo daily for 7 days
  6 additional subjects will receive 300 mg NYX-2925 daily for 7 days and undergo lumbar puncture on Day 6 in order to have two CSF samples taken (CSF Cohort).
  Interventions: Drug: NYX-2925

INTERVENTIONS:
Drug: NYX-2925 — NYX-2925 is a small molecule that acts as an N-methyl-D-aspartate receptor (NMDAR) functional glycine-site partial agonist.

SUMMARY:
This is a first in human study of NYX-2925. It will evaluate single and multiple ascending doses of NYX-2925 in healthy volunteers.

DETAILED DESCRIPTION:
This is a first in human study of NYX-2925. This is a randomized, double-blind, sponsor-open, placebo-controlled, single and multiple ascending dose, parallel safety, tolerability, and PK study of oral NYX-2925 in healthy volunteers. The single ascending dose phase will comprise up to five dose groups. There will be up to 3 dose groups in the multiple ascending dose phase. One open-label dose group will be repeated in the multiple ascending dose phase to collect cerebrospinal fluid (CSF) samples, in order to explore central nervous system penetration. One elderly cohort (single dose) will be completed after all single and multiple dose escalation groups have completed. One open-label dose group will be repeated in the single ascending dose phase to collect CSF samples, in order to establish a more complete cerebral spinal fluid pharmacokinetic profile.

The influence of food ("food effect") on the bioavailability and pharmacokinetics of NYX-2925 will be explored in one dose group in the single ascending dose phase.

A data review committee will review safety and tolerability (adverse events and other relevant data), plus preliminary pharmacokinetic data, prior to proceeding to the next higher dose group, cohort, and/or phase of the study, as well as administration of the fed dose in the food effect group.

Stopping rules for individual study participants and dose groups or cohorts are established in order to evaluate the dose escalation scheme, the need to stop or terminate dosing, or to establish the maximum tolerated dose. If a cohort is stopped due to safety or tolerability concerns, the previous cohort may be repeated to determine the highest tolerated dose.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects.
2. 18 to 55 years of age, inclusive, at the time of signing the informed consent form (ICF). 55 to 80 years of age for elderly cohort.
3. Female subjects with a negative serum pregnancy test prior to entry into the study and who are practicing an adequate method of birth control (e.g., oral or parenteral contraceptives, intrauterine device, barrier, abstinence) and who do not plan to become pregnant during the course of the study.
4. Male subjects and their female sexual partner should use an acceptable method of birth control during the study. Male subjects must agree to use barrier contraception (condom with spermicide), and refrain from sperm donation, from the first dose of study drug until 90 days after the last dose of study drug.
5. Clinical laboratory values within normal limits or deemed not clinically significant by the investigator and/or the sponsor.
6. Ability to understand the requirements of the study, provide written informed consent, abide by the study restrictions, and agree to return for the required assessments.
7. Subject is judged to be in good health as determined by the investigator based on the results of a medical history, physical examination (PE), clinical laboratory profile, and electrocardiogram (ECG) performed during the screening period and confirmed prior to dosing.
8. Body mass index (BMI) between 18 and 30 kg/m2 (inclusive).
9. Normal renal and hepatic function, with calculated creatinine clearance ≥ 90 mL/minute (Cockcroft-Gault Formula) at Screening or ≥ 60 mL/minute only in the case of the elderly cohort.

Exclusion Criteria:

1. Clinically significant alcohol or other substance abuse within the last 24 months, in the opinion of the investigator; or, unable to abstain from alcoholic beverages during the course of the study.
2. Positive screen for alcohol or drugs of abuse (with the exception of a positive result considered by the investigator to be directly attributable to prescription medication approved for subject use): including benzodiazepines, opiates, cocaine, cannabinoids, and amphetamines.
3. History of smoking or tobacco use within 30 days of Screening.
4. Women who are pregnant, breast feeding, or planning to become pregnant during the course of the study.
5. History of allergy, sensitivity, or intolerance to NMDAR ligands including ketamine, dextromethorphan, memantine, methadone, dextropropoxyphene, or ketobemidone, as well as current use of such agents.
6. Received an investigational drug or device within 30 days (or 5 half-lives, whichever is longer) of dosing.
7. Previously assigned to treatment during this study (except those who did not take study medication).
8. Screening QT interval corrected for heart rate by Fridericia's formula (QTcF) > 450 (males) or 470 (females) millisecond (msec) or an ECG that is not suitable for QT measurements (e.g., poorly defined termination of T-wave in the investigator's opinion).
9. Type I or Type II diabetes.
10. History of severe renal or hepatic impairment, in the opinion of the investigator or the sponsor-designated medical monitor.
11. History of excessive bleeding, blood thinners within 6 months, antibiotics or infection within 3 months (CSF cohort only), lumbar spine abnormality, history of elevated intracranial pressure, normal pressure hydrocephalus or other neurological conditions considered clinically significant by the investigator.
12. Human immunodeficiency virus infection, hepatitis, or other ongoing infectious disease that the investigator considers clinically significant.
13. Current evidence of dysplasia or history of malignancy (including lymphoma and leukemia) in the last 5 years, with the exception of successfully treated non-metastatic basal cell or squamous cell carcinoma of the skin or localized carcinoma in situ of the cervix.
14. History of seizures.
15. History of gastrointestinal disease or surgery (except simple appendectomy or hernia repair), which can influence the absorption of the study drug.
16. History of any type of psychosis (including but not limited to bipolar disease or schizophrenia).
17. Medical history or conditions that, in the opinion of the investigator, would preclude safe study participation, or interfere with study procedures/assessments.
18. Evidence of an infection at the time of clinic admission, in the opinion of the investigator.
19. Poor venous access.
20. Use of prescription or over-the-counter medications, including herbal therapies within 7 days prior to dosing, or during the treatment and follow-up periods. Use of St. John's wort within 14 days prior to dosing, or during the treatment and follow-up periods. Occasional aspirin may be used at the investigator's discretion.
21. Unable to eat a standardized meal offered by the study center.
22. Donated or had a loss of blood or plasma within 8 weeks prior to dosing.
23. Grapefruit juice or Seville oranges within 14 days prior to dosing or during the dosing period.
24. Heart rate ≤ 45 beats per minutes.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2016-07; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events | Subjects will be followed for up to 30 days post-dose

SECONDARY OUTCOMES:
Cmax of NYX-2925 | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose
Tmax of NYX-2925 | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose
AUC of NYX-2925 | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose
Half-life of NYX-2925 | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose
Clearance of NYX-2925 | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose
Volume of distribution of NYX-2925 | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose
Renal elimination of NYX-2925 | 0-4, 4-8, 8-12, 12-16, and 16-24 hours post dose.
Food effect of NYX-2925 following consumption of a high-fat, high-caloric meal | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose
CSF penetration of NYX-2925 in CSF cohort | 1, 2, 2.5, and 8 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Sanabria, MD, Principal Investigator — Spaulding Clinical Research LLC; Laurel Sindelar, Study Director — Aptinyx Inc.
Locations (1):
- Spaulding Clinical, West Bend, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes